CLINICAL TRIAL: NCT03064087
Title: Validation of Human Papillomavirus Assays and Collection Devices for HPV Testing on Self-samples and First-void Urine Samples (VALHUDES)
Brief Title: Validation of Human Papillomavirus Assays and Collection Devices for Self-samples and Urine Samples
Acronym: VALHUDES
Status: Active, not recruiting | Type: Observational
Sponsor: Marc Arbyn (Other Government)
Collaborators: Algemeen Medisch Laboratorium (Unknown); Universiteit Antwerpen (Other); Regionaal Ziekenhuis Heilig Hart Tienen (Other); University Hospital, Antwerp (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor-Investigator, Marc Arbyn, Coordinator Unit Cancer Epidemiology (Belgian Cancer Centre), Sciensano
Organization: Sciensano (Other Government)
Other Study IDs: WIV-ISP_2017_001
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3
Keywords: Self-Sampling; HPV Testing; Diagnostic Test Accuracy; Cervical Intraepithelial Neoplasia; Urine; Cervical Cancer Screening
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — First-void urine sample, vaginal self-sample and cervical cell sample collected by a gynecologist. No human DNA is extracted from the samples but the samples can contain HPV DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Colli-Pee — First, two first-void urine samples will be collected with the Colli-Pee device (Novosanis NV, Wijnegem, Belgium) at home, the day before a visit to the colposcopy centre at a gynecology clinic.
Device: Multi-Collect Swab — At the colposcopy clinic, one vaginal self-sample will be collected with the Multi-Collect Swab (Abbott GmbH & Co. KG, Wiesbaden, Germany).
Device: Evalyn Brush — Another vaginal self-sample will be collected also at the colposcopy centre either with the Evalyn Brush (Rovers Medical Devices B.V., Oss, Netherlands)
Device: Qvintip — or with Qvintip (Aprovix AB, Uppsala, Sweden).
Diagnostic Test: Abbott RealTime High Risk HPV — The hrHPV assay used, will be the Abbott PCR (Abbott GmbH & Co. KG, Wiesbaden, Germany), which detects separately DNA of HPV16 and HPV18, as well as the pool of twelve other hrHPV types (HPV 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68). The accuracy of this PCR assay for the detection of CIN2+ will be determined on all samples: on the first urine sample and on the vaginal and cervical samples. Furthermore, it is possible that in the future other assays will be validated.

SUMMARY:
The VALHUDES study is a Diagnostic Test Accuracy study that aims to document the clinical accuracy of hrHPV testing on urine samples, collected under standardised and optimised conditions, and on two types of vaginal self-samples and compare results with those from matching samples taken by a clinician.

DETAILED DESCRIPTION:
The samples are collected from patients referred to colposcopy because of prior cervical abnormalities. The patient takes at home two urine samples with the Colli-Pee device (a device that allows to collect first-void urine), the day before the visit to the colposcopy centre. At the colposcopy centre, two vaginal self-samples are taken by the patient herself: one with a cotton swab and a second with a plastic brush. Finally, the gynecologist takes a cervical Pap smear with a Cervex-Brush Combi.

A real-time PCR test will be used to detect DNA of high-risk HPV types. It is possible that in the future also other tests will be validated on these samples. The colposcopy and histological findings will be used as the gold standard. The main purpose of the study is to assess the relative diagnostic tests accuracy of hrHPV testing on self- and urine samples compared to hrHPV testing on cervical samples taken by a clinician. Furthermore, the participating women will receive also a questionnaire which can give insights into the attitudes and preferences of the women with regard to the self-sampling devices.

ELIGIBILITY:
Inclusion Criteria:

* Women with previous abnormal cervical cancer screening test results
* Women between the ages of 25 and 64

Exclusion Criteria:

* Hysterectomised women
* Women with known pregnancy
* Non-consenting women
* Women that are not able to understand and to sign the informed consent

Ages: 25 Years to 64 Years | Sex: Female
Age Groups: Adult
Study Population: 500 women referred to a participating Belgian colposcopy centre (University Hospital of Ghent, Brussels and Antwerp, Hospital of Tienen) because of a previous abnormal cervical cancer screening test result, will be enrolled after obtaining informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-11-17 (Estimated)

PRIMARY OUTCOMES:
Clinical accuracy | up to 18 months
  • Relative sensitivity and specificity of hrHPV testing on first-void urine vs clinician-collected samples.
Clinical accuracy | up to 18 months
  • Relative sensitivity and specificity of hrHPV testing on vaginal self-samples vs clinician-collected samples.

SECONDARY OUTCOMES:
Clinical accuracy | up to 18 months
  • Absolute sensitivity and specificity for finding underlying CIN2+ of hrHPV testing on urine, self- and clinician-collected samples.
Clinical accuracy | up to 18 months
  • Relative sensitivity and specificity of hrHPV testing on samples taken with the Qvintip vs the Evalyn Brush (non-matched comparison) and on urine samples vs the different vaginal self-samples (matched comparison)
Clinical accuracy | up to 18 months
  • An intermediate statistical analysis will be performed after that 100 patients are included to verify whether all processes run as expected. Possible protocol adjustments may be considered after this intermediate analysis.
Analytical performance | up to 18 months
  • Concordance of the presence of hrHPV and of the partial HPV genotyping results applied on urine, self- and clinician-collected samples; correlation in viral load (expressed as cycle number values) between samples.
Analytical performance | up to 18 months
  • Positivity rates for beta-globin in the different types of samples.
Analytical performance | up to 18 months
  • Correlation of cycle number values for HPV16, HPV18, other hrHPV and beta-globin between the different types of samples.
Acceptance and preferences | up to 18 months
  • Acceptance of self-sampling, preferences of women (assessed from a questionnaire and from participation rate [number of women who participate/number of women approached]).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Arbyn, PhD, Principal Investigator — Unit of Cancer Epidemiology, Belgian Cancer Centre, Sciensano
Locations (5):
- Belgium (5):
  - UZ Brussels, Brussels, Brussels Capital
  - UZ Ghent, Ghent, East Flanders
  - Heilig Hart Ziekenhuis Tienen, Tienen, Flemish Brabant
  - UZ Antwerp, Antwerp
  - Centre Hospitalier Universitaire de Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Background] Arbyn M, Snijders PJ, Meijer CJ, Berkhof J, Cuschieri K, Kocjan BJ, Poljak M. Which high-risk HPV assays fulfil criteria for use in primary cervical cancer screening? Clin Microbiol Infect. 2015 Sep;21(9):817-26. doi: 10.1016/j.cmi.2015.04.015. Epub 2015 May 1. PMID 25936581
- [Background] Arbyn M, Castle PE. Offering Self-Sampling Kits for HPV Testing to Reach Women Who Do Not Attend in the Regular Cervical Cancer Screening Program. Cancer Epidemiol Biomarkers Prev. 2015 May;24(5):769-72. doi: 10.1158/1055-9965.EPI-14-1417. Epub 2015 Feb 24. PMID 25713024
- [Background] Verdoodt F, Jentschke M, Hillemanns P, Racey CS, Snijders PJ, Arbyn M. Reaching women who do not participate in the regular cervical cancer screening programme by offering self-sampling kits: a systematic review and meta-analysis of randomised trials. Eur J Cancer. 2015 Nov;51(16):2375-85. doi: 10.1016/j.ejca.2015.07.006. Epub 2015 Aug 18. PMID 26296294
- [Background] Vorsters A, Van den Bergh J, Micalessi I, Biesmans S, Bogers J, Hens A, De Coster I, Ieven M, Van Damme P. Optimization of HPV DNA detection in urine by improving collection, storage, and extraction. Eur J Clin Microbiol Infect Dis. 2014 Nov;33(11):2005-14. doi: 10.1007/s10096-014-2147-2. Epub 2014 Jun 12. PMID 24916950
- [Derived] Van Keer S, Latsuzbaia A, Vanden Broeck D, De Sutter P, Donders G, Doyen J, Tjalma WAA, Weyers S, Arbyn M, Vorsters A. Analytical and clinical performance of extended HPV genotyping with BD Onclarity HPV Assay in home-collected first-void urine: A diagnostic test accuracy study. J Clin Virol. 2022 Oct;155:105271. doi: 10.1016/j.jcv.2022.105271. Epub 2022 Aug 24. PMID 36049283
- [Derived] Latsuzbaia A, Vanden Broeck D, Van Keer S, Weyers S, Tjalma WAA, Doyen J, Donders G, De Sutter P, Vorsters A, Peeters E, Arbyn M. Clinical Performance of the RealTime High Risk HPV Assay on Self-Collected Vaginal Samples within the VALHUDES Framework. Microbiol Spectr. 2022 Oct 26;10(5):e0163122. doi: 10.1128/spectrum.01631-22. Epub 2022 Sep 1. PMID 36047900
- [Derived] De Pauw H, Donders G, Weyers S, De Sutter P, Doyen J, Tjalma WAA, Vanden Broeck D, Peeters E, Van Keer S, Vorsters A, Arbyn M. Cervical cancer screening using HPV tests on self-samples: attitudes and preferences of women participating in the VALHUDES study. Arch Public Health. 2021 Aug 30;79(1):155. doi: 10.1186/s13690-021-00667-4. PMID 34462004
- [Derived] Arbyn M, Peeters E, Benoy I, Vanden Broeck D, Bogers J, De Sutter P, Donders G, Tjalma W, Weyers S, Cuschieri K, Poljak M, Bonde J, Cocuzza C, Zhao FH, Van Keer S, Vorsters A. VALHUDES: A protocol for validation of human papillomavirus assays and collection devices for HPV testing on self-samples and urine samples. J Clin Virol. 2018 Oct;107:52-56. doi: 10.1016/j.jcv.2018.08.006. Epub 2018 Aug 22. PMID 30195193